CLINICAL TRIAL: NCT04574557
Title: Hepatic Micro RNA Expression In Non Alcoholic Fatty Liver Disease
Brief Title: Micro RNA Levels in NAFLD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nourhan Mahmoud Abbas, Assistant lecturer at tropical medicine and gastroenterology department, Assiut University
Other Study IDs: micro RNA in NAFLD
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: micro RNA
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — miRNA was isolated from serum using a miRNeasy Mini Kit (Qiagen, Cat; 217004) cDNA was isolated from obtained miRNA samples using a miScript Reverse Transcription Kit (Qiagen, Cat; 218060) Quantitative Real-Time PCR (qPCR) will be done using (miScript SYBR Green PCR Kit Qiagen Cat. No: 218073)The qPCR assays were performed in duplicate The relative expressions of Three miRNAs were selected for RT-PCR validation Two were selected from over-expressed miRNAs (miR-34a, miR-146b), one from under-expressed miRNAs (miR-122) were analyzed using the standard 2-ΔΔCT method. These miRNAs were selected due to their pathophysiological relation with NASH.
  Predicted gene targets of all differentially expressed miRNAs will be identified. Genes with functions that are potentially relevant to the pathogenesis of NASH and gene targets that are commonly studied e.g. lipogenesis (e.g. FAS), inflammation (c-JUN kinase) will be included in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: micro RNA — miRNA was isolated from serum using a miRNeasy Mini Kit (Qiagen, Cat; 217004)cDNA was isolated from obtained miRNA samples using a miScript Reverse Transcription Kit (Qiagen, Cat; 218060) Quantitative Real-Time PCR (qPCR) will be done using (miScript SYBR Green PCR Kit Qiagen Cat. No: 218073)The qPCR assays were performed in duplicate The relative expressions of Three miRNAs were selected for RT-PCR validation Two were selected from over-expressed miRNAs (miR-34a, miR-146b), one from under-expressed miRNAs (miR-122) were analyzed using the standard 2-ΔΔCT method. These miRNAs were selected due to their pathophysiological relation with NASH.
  Predicted gene targets of all differentially expressed miRNAs will be identified. Genes with functions that are potentially relevant to the pathogenesis of NASH and gene targets that are commonly studied e.g. lipogenesis (e.g. FAS), inflammation (c-JUN kinase) will be included in the study

SUMMARY:
* Epidemiological study of NAFLD, NASH patients.
* Descriptions of altered miRNA profiles in NAFLD patients especially with fibrosis. - Explore the role of circulating miRNAs as biomarkers for the early diagnosis and evaluation of NAFLD patient with fibrosis.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is defined as the presence of hepatic steatosis (>5%-10% of hepatocytes are fatty) in people without history of excessive alcohol consumption (>21 drinks/week in men and > 14drinks/week in women) and other disease etiologies that result in fatty liver.

The presence of coexisting risk factors such as diabetes, metabolic syndrome, and obesity increases the risk of NAFLD. As a consequence of obesity pandemic and type 2 diabetes, an increased number of patients with NASH-the most severe form of NAFLD-is expected in the near future.

According to the latest epidemiological studies, the prevalence of NAFLD is approximately 25% worldwide.

In developed countries such as the United States, the prevalence of NAFLD is 30%. In developing countries such as China, the prevalence has reached up to 32.9%.

NAFLD comprises a spectrum of pathological conditions, Including simple steatosis (NAFL), nonalcoholic steatohepatitis (NASH), fibrosis, cirrhosis and hepatocellular carcinoma (HCC).

Studies have shown that approximately one-sixth of NAFL patients progress to NASH, and 20% of NASH patients can develop cirrhosis.

The traditional view suggests that HCC formation is a multi-stage process, involving inflammation, fibrosis and cirrhosis. However, recent research found that NASH can progress to HCC without fibrosis and cirrhosis.

NAFLD patients are often associated with higher risk of developing both cardiovascular disease and type 2diabetes, therefore early diagnosis of NAFLD and intervention would greatly benefit the patient by preventing the progression of major hepatic and extra hepatic manifestations.

In patients with NAFLD, the most important factor is the assessment of fibrosis severity and monitoring fibrosis progression. Most patients remain asymptomatic until their liver functionis compromised.

Thus, the identification of the presence and severity of liver fibrosis remains a clinical challenge.

Therefore, early predictors need to be investigated.

Multiple factors are involved in NAFLD development, including lipotoxicity, insulin resistance, endoplasmic reticulum stress, adipose tissue, gut microbiota, and genetics [9].

Our understanding of the pathogenesis of this disease remains limited because of its broad range and complexity.

Liver biopsy is the current gold standard in diagnosis and prognosis; nevertheless, it is an expensive and invasive procedure with high sampling error and risk of complications including pain bleeding; and, in very rare cases, death.

A biomarker is a patient characteristic assessed as an indicator of a normal or a pathologic process or of a biological response to treatment.

Unfortunately, to date, existing non- or minimally invasive biomarkers are inadequate.

Circulating extracellular vesicles (exosomes and ectosomes) contain various cellular molecules such as proteins, mRNA, miRNAs, and DNA can serve as biomarkers in NAFLD and NASH.

MicroRNAs (miRNAs) are short, non-coding single stranded RNAs strand of 20-25 nucleotides. miRNAs play complicated and important roles in regulating the expression of downstream genes .

MiRNAs contribute to the pathogenesis of NAFLD/NASH at various levels of disease development and progression and probably are the most extensively studied epigenetic modifications in NAFLD .

miR-122 is the most abundant miRNA in human liver, representing more than 70% of the total liver miRNA pool.

During hepatocytes maturation, miR-122 stimulates the expression of 24 hepatocytes-specific genes, including hepatocyte nuclear factor 6 (HNF6) [13], and in liver regeneration it has been reported to regulate hepatocytes proliferation and differentiation, recapitulating the developmental processes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Elevated aminotransferases
3. Ultrasonographic presence of hyper echogenic liver
4. fibroscan with a diagnosis of non-alcoholic fatty liver disease with fibrosis (NASH) without cirrhosis done no more than 6 months before the study.

Exclusion Criteria:

1. A history of any level of alcohol consumption
2. Any other form of chronic liver disease
3. Use of any medications thought to cause or affect NAFLD
4. Acute or chronic infection
5. History of cancer
6. Chronic kidney diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a hospital-based study will carried out prospectively in Tropical Medicine and Gastroenterology Department, Al-Rajhi Liver Hospital, Assiut University.
  Based on determining the main outcome variable, the estimated minimum required sample size is 80 patients (40 in each group cases and control).
  cases : 40 patients of NAFLD patients with the previus eligibility criteria A control group : of 40 healthy age and sex-matched subjects with normal liver enzymes and abdominal ultrasonography findings
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Descriptions of altered miRNA profiles in NAFLD patients especially with fibrosis. | baseline
  Explore the role of circulating miRNAs as biomarkers for the early diagnosis and evaluation of NAFLD patient with fibrosis

REFERENCES:
- [Background] Dodds WJ, Hogan WJ, Miller WN. Reflux esophagitis. Am J Dig Dis. 1976 Jan;21(1):49-67. doi: 10.1007/BF01074140. No abstract available. PMID 3966
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Cotter TG, Rinella M. Nonalcoholic Fatty Liver Disease 2020: The State of the Disease. Gastroenterology. 2020 May;158(7):1851-1864. doi: 10.1053/j.gastro.2020.01.052. Epub 2020 Feb 13. PMID 32061595
- [Background] Zhou J, Zhou F, Wang W, Zhang XJ, Ji YX, Zhang P, She ZG, Zhu L, Cai J, Li H. Epidemiological Features of NAFLD From 1999 to 2018 in China. Hepatology. 2020 May;71(5):1851-1864. doi: 10.1002/hep.31150. PMID 32012320
- [Background] Adams LA, Lymp JF, St Sauver J, Sanderson SO, Lindor KD, Feldstein A, Angulo P. The natural history of nonalcoholic fatty liver disease: a population-based cohort study. Gastroenterology. 2005 Jul;129(1):113-21. doi: 10.1053/j.gastro.2005.04.014. PMID 16012941
- [Background] Febbraio MA, Reibe S, Shalapour S, Ooi GJ, Watt MJ, Karin M. Preclinical Models for Studying NASH-Driven HCC: How Useful Are They? Cell Metab. 2019 Jan 8;29(1):18-26. doi: 10.1016/j.cmet.2018.10.012. Epub 2018 Nov 15. PMID 30449681
- [Background] Baffy G, Brunt EM, Caldwell SH. Hepatocellular carcinoma in non-alcoholic fatty liver disease: an emerging menace. J Hepatol. 2012 Jun;56(6):1384-91. doi: 10.1016/j.jhep.2011.10.027. Epub 2012 Feb 9. PMID 22326465
- [Background] Anstee QM, Targher G, Day CP. Progression of NAFLD to diabetes mellitus, cardiovascular disease or cirrhosis. Nat Rev Gastroenterol Hepatol. 2013 Jun;10(6):330-44. doi: 10.1038/nrgastro.2013.41. Epub 2013 Mar 19. PMID 23507799
- [Background] Baranova A, Younossi ZM. The future is around the corner: Noninvasive diagnosis of progressive nonalcoholic steatohepatitis. Hepatology. 2008 Feb;47(2):373-5. doi: 10.1002/hep.22140. No abstract available. PMID 18220279
- [Background] Than NN, Newsome PN. A concise review of non-alcoholic fatty liver disease. Atherosclerosis. 2015 Mar;239(1):192-202. doi: 10.1016/j.atherosclerosis.2015.01.001. Epub 2015 Jan 13. PMID 25617860
- [Background] Malhi H. Emerging role of extracellular vesicles in liver diseases. Am J Physiol Gastrointest Liver Physiol. 2019 Nov 1;317(5):G739-G749. doi: 10.1152/ajpgi.00183.2019. Epub 2019 Sep 23. PMID 31545919
- [Background] Xiao G, Zhu S, Xiao X, Yan L, Yang J, Wu G. Comparison of laboratory tests, ultrasound, or magnetic resonance elastography to detect fibrosis in patients with nonalcoholic fatty liver disease: A meta-analysis. Hepatology. 2017 Nov;66(5):1486-1501. doi: 10.1002/hep.29302. Epub 2017 Sep 26. PMID 28586172
- [Background] Pu K, Wang Y, Bai S, Wei H, Zhou Y, Fan J, Qiao L. Diagnostic accuracy of controlled attenuation parameter (CAP) as a non-invasive test for steatosis in suspected non-alcoholic fatty liver disease: a systematic review and meta-analysis. BMC Gastroenterol. 2019 Apr 8;19(1):51. doi: 10.1186/s12876-019-0961-9. PMID 30961539